CLINICAL TRIAL: NCT06975839
Title: Evaluate the Efficacy of Local Metformin Gel Application Following Surgical Removal of Mandibular Third Molar
Brief Title: Local Metformin Gel and Impacted Lower Third Molar
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Shaimaa Mohsen, associate professor, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 8
Record Dates: First submitted 2025-05-09; First posted 2025-05-16 (Actual); Last update posted 2025-05-16 (Actual); Status verified 2025-05

CONDITIONS: Impacted Third Molar Tooth
MeSH Terms: interventions — Metformin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- metformin (Experimental)
  Interventions: Drug: Metformin
- non metformin (Active Comparator)
  Interventions: Drug: non metformin gel

INTERVENTIONS:
Drug: Metformin — local application of metformin gel after surgical removal of lower third molar tooth
  Arms: metformin
Drug: non metformin gel — local application of placebo gel after surgical removal of lower third molar tooth
  Arms: non metformin

SUMMARY:
* Completed medical and dental history will take for all patients and the position of the impacted teeth will evaluate by panoramic films. Patients will fully inform about the treatment procedures, follow-up examinations and complications of surgical procedures.
* The study will be carried out as a randomized controlled clinical trial. Randomly, by the use of predefined computer-generated randomization table, the eligible patients will be randomized in equal proportions between Study group: patients will receive 1% Metformin gel in the socket following removal of the impacted third molar and Control group: patients will receive placebo gel 2% hydroxymethyl cellulose.All surgeries will be performed under complete aseptic conditions. Before surgery, the patient's mouth will be rinsed with a chlorhexidine digluconate solution 0.2% for 2 minutes. Surgery will carry out under local anesthesia consisting of 4% articain hydrochloride with 1:100,000 adrenaline.
* Full thickness mucoperiosteal flap will be raised to expose sufficient bone on lateral and distal aspect of the impacted molar. Removal of bone will be done with stainless steel bur under Constant irrigation with normal saline while removing bone to prevent thermal necrosis.
* When necessary, sectioning of crown and roots will be performed with a fissure bur. After tooth extraction, the alveolus will be inspected, curetted, and irrigated with 0.9% sterile saline solution.
* Surgical removal of impacted mandibular third molar will be done,1% metformin gel or placebo gel in the socket following removal of the impacted third molar .
* The mucoperiosteal flap will be repositioned and sutured with 3-0 black silk suture.

ELIGIBILITY:
Inclusion Criteria:

* • Age ≥18ys

  * no systemic disease
  * impacted mandibular third molar class II position B on Pell- Gregory classification

Exclusion Criteria:

* • history of metabolic or systemic diseases affecting bone or healing process,

  * local infection,
  * tobacco use,
  * oral contraceptive,
  * pregnancy and lactation
  * patients who had taken analgesics or anti-inflammatories for 1 week prior to enrollment in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-02-01 (Estimated)

PRIMARY OUTCOMES:
bone dentisty | 6months
  by CBCT